CLINICAL TRIAL: NCT05096806
Title: Effects of Semi-standarized Acupuncture in Chronical Symptomatic Osteoarthritis of the Knee Through: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat de Girona (Other)
Responsible Party: Principal Investigator, Tomás Tegiacchi, Principal Investigator, Universitat de Girona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBRU0021-21
Record Dates: First submitted 2021-09-29; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Acupuncture; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care plus TENS (Active Comparator): Participants in this group will receive transcutaneous electrical nerve stimulation (TENS) and usual care.
  TENS treatment will perform in the region of the knee and the extensor muscles for 20 minutes, 2 times a week. 4 electrodes will be placed, 2 on the proximal region of the internal and external vastus, and the other 2 on the distal region of the motor plate.
  Usual care will consist in home exercises with toning exercises of the extensor apparatus, pelvic region and musculoskeletal stretching exercises of 2 weekly sessions, the recommendation of daily activity of walking for 1 hour daily as an active lifestyle and the recommendation of the reduction of body weight in the case of being above normal weight. There will be a total of 6 face-to-face sessions at the rate of 2 weekly sessions
  Interventions: Device: TENS
- Usual care plus Acupuncture (Experimental): Participants in this group will receive acupuncture treatment and usual care.
  Acupuncture treatment will consist in 20-minute semi-standardized acupuncture sessions, 2 times a week. The intervention will consist of the insertion of 8 needles: 4 in points located in the knee (points St34, St35, XiYan and Sp10) and 4 more sensitive to palpation points located between the knee and the ankle. Stimulation will be performed to obtain local spasm response, the needles will be left for 20 minutes and then removed. The needles will be sterile disposable silicone needles of 0.20x20mm and 0.20x40mm.
  Usual care will be the same described in the Usual care plus TENS group
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a non-pharmacological technique that consists in the stimulation of specific points located in the skin surface. Points are stimulated by piercing the skin with fine needles.
  Arms: Usual care plus Acupuncture
Device: TENS — TENS is a therapy that uses low voltage electrical current to provide pain relief. A TENS unit consists of a battery-powered device that delivers electrical impulses through electrodes placed on the surface of your skin. The electrodes are placed at or near nerves where the pain is located or at trigger points.
  Other Names: Transcutaneous electrical nerve stimulation
  Arms: Usual care plus TENS

SUMMARY:
Introduction:

Knee osteoarthritis is a long-term rheumatic disease with a significant impact on the patient's quality of life and the socio-economic development of societies. The usual treatment consists of non-steroidal anti-inflammatory drugs as a palliative measure. The decrease in the beneficial effect and the appearance of serious long-term adverse effects make it necessary to look for other therapeutic procedures. Acupuncture is a non-pharmacological treatment that could reduce pain and improve functionality in this condition, however current scientific evidence is limited. A previous study has observed a clinical improvement in the combination of sensitized local and peripheral points in the treatment of knee osteoarthritis but studies with a larger sample are needed to confirm these results.

Objective:

Assess the effectiveness of acupuncture using a combination of local and peripheral sensitized points in the treatment of active knee osteoarthritis.

Methods:

A randomized clinical trial will be performed in a hospital centre with 2 groups. The control group will standard treatment plus transcutaneous electrical nerve stimulation, while the intervention group will receive acupuncture in addition to standard care. Study outcomes will be pain, quality of life, function, exercise adherence, drug intake, adverse effects, and body mass index. There will be a 12-month post-intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Usual painful episode of 3 months or more
* Morning stiffness of 15 minutes or more
* Pain equal to or greater than 5 on the VAS
* Grade 2 or greater on the Kellgren-Lawrence scale

Exclusion Criteria:

* Corticosteroid infiltration in the 3 months prior to recruitment
* Rehabilitation treatment one month prior to recruitment
* With a knee prosthesis
* Needle phobia
* Pregnancy
* With pacemakers
* Cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain at post intervention | At the end of the intervention, at the 4th week of the study
  Pain will be assessed using the visual analogue scale (VAS)
Change from Baseline Knee function at postintervention | At the end of the intervention, at the 4th week of the study
  Knee function will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Change from Baseline Quality of life at postintervention | At the end of the intervention, at the 4th week of the study
  Quality of life will be assessed using the SF-12 questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

SECONDARY OUTCOMES:
Change from Baseline Pain at 4 months | 16 weeks afther the end of the intervention, at the 20th week of the study
  Pain will be assessed using the visual analogue scale (VAS)
Change from Baseline Knee function at 4 months | 16 weeks afther the end of the intervention, at the 20th week of the study
  Knee function will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Change from Baseline Quality of life at 4 months | 16 weeks afther the end of the intervention, at the 20th week of the study
  Quality of life will be assessed using the SF-12 questionnaire. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Drug intake postintervention | through study completion, an average of 1 year
  Rescue drug intake will be collected in the data collection notebooks
Adverse events postintervention | through study completion, an average of 1 year
  Any adverse event related with the treatments will be will be noted in a collection sheet.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roos EM, Arden NK. Strategies for the prevention of knee osteoarthritis. Nat Rev Rheumatol. 2016 Feb;12(2):92-101. doi: 10.1038/nrrheum.2015.135. Epub 2015 Oct 6. PMID 26439406
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] Woods B, Manca A, Weatherly H, Saramago P, Sideris E, Giannopoulou C, Rice S, Corbett M, Vickers A, Bowes M, MacPherson H, Sculpher M. Cost-effectiveness of adjunct non-pharmacological interventions for osteoarthritis of the knee. PLoS One. 2017 Mar 7;12(3):e0172749. doi: 10.1371/journal.pone.0172749. eCollection 2017. PMID 28267751
- [Background] Cao H, Bourchier S, Liu J. Does Syndrome Differentiation Matter? A Meta-Analysis of Randomized Controlled Trials in Cochrane Reviews of Acupuncture. Med Acupunct. 2012 Jun;24(2):68-76. doi: 10.1089/acu.2011.0846. PMID 24761164
- [Background] Li J, Li YX, Luo LJ, Ye J, Zhong DL, Xiao QW, Zheng H, Geng CM, Jin RJ, Liang FR. The effectiveness and safety of acupuncture for knee osteoarthritis: An overview of systematic reviews. Medicine (Baltimore). 2019 Jul;98(28):e16301. doi: 10.1097/MD.0000000000016301. PMID 31305415